CLINICAL TRIAL: NCT06517823
Title: Efficacy and Safety of the Fixed-Dose Combination of Etoricoxib/Cyanocobalamin Versus Etoricoxib in the Treatment of Patients with Acute Low Back Pain
Brief Title: Efficacy and Safety of Etoricoxib/Cyanocobalamin Versus Etoricoxib for Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30952-III-23(1)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Low-back Pain
Keywords: Acute Low -back Pain; Acute pain; Etoricoxib; Cyanocobalamin
MeSH Terms: conditions — Acute Pain | interventions — Etoricoxib; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etoricoxib+Cyanocobalamin (Experimental): Administered orally, 1 tablet a day for 7 days.
  Interventions: Drug: Etoricoxib + Cyanocobalamin fixed dose
- Etoricoxib (Active Comparator): Administered orally, 1 pill a day for 7 days.
  Interventions: Drug: Etoricoxib fixed dose

INTERVENTIONS:
Drug: Etoricoxib + Cyanocobalamin fixed dose — One tablet of 90 mg / 0.50 mg a day
  Other Names: Etori + Cyano
  Arms: Etoricoxib+Cyanocobalamin
Drug: Etoricoxib fixed dose — One pill of 90 mg a day
  Other Names: Etori
  Arms: Etoricoxib

SUMMARY:
Phase III longitudinal, multicenter, randomized, double-blind clinical trial. The aim of this study is to evaluate the efficacy and safety of the Fixed-Dose Combination of Etoricoxib/Cyanocobalamin Versus Etoricoxib in Patients With Acute Low Back Pain

DETAILED DESCRIPTION:
Researchers will compare the fixed-dose combination of Etoricoxib/Cyanocobalamin versus Etoricoxib in acute low back pain by comparing the proportion of patients that reported an improvement in pain during the 7 days of follow up. The adverse events related to the interventions will be registered during follow up.

Participants will:

* Be randomized into one of the 2 intervention groups (A or B)
* Visit the clinic in 3 occasions (day 0, day 3 of follow up and day 7 of follow up)
* In case needed the patient could take 50 mg of tramadol, as a rescue medication, previous authorization of de principal investigator

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study and give written informed consent
* Patient with pain reported as moderate to severe intensity with ≥ 40 mm on the Visual Analog Scale (VAS).
* At least 4 points on the "Douleur Neuropathique-4 items" (DN-4) scale.
* Diagnosis of acute low back pain as a first-time episode or a previous episode 6 months before the enrollment day and lasting no more than 6 weeks.
* Women of childbearing potential under a medically acceptable method of contraception

Exclusion Criteria:

* Patients participating in another clinical trial involving an investigational treatment or participation in one within 4 weeks prior to study start
* Patients in whom the participation in the study may be influenced (employment relationship with the research site or sponsor, inmates, etc.)
* At medical discretion, a disease that affects prognosis and prevents outpatient management, for example, but not limited to: end-stage cancer, kidney, heart, respiratory or liver failure, mental illness or with scheduled surgical or hospital procedures
* History/presence of any disease or condition that, in the opinion of the Investigator, could pose a risk for the patient or confusing the efficacy and safety of the investigational product
* Patients in whom the study drug is contraindicated for medical reasons
* Patients with allergy or hypersensitivity to the active substance of the study drugs, related products or excipients (Etoricoxib of Cyanocobalamin)
* Pregnant women, women breastfeeding or planning a pregnancy during the conducting the study
* Significant history of gastrointestinal diseases (e.g., gastric ulcer, Crohn's disease, Ulcerative Colitis, etc.)
* Active opioid and/or NSAID treatment including COX-2 inhibitors, reported in the medical record within the last 72 hours of study entry.
* Patients with a history of congestive heart failure: NYHA II-IV.
* Concomitant use of strong CYP1A2 inhibitors (e.g., fluvoxamine, ciprofloxacin, etc.).
* Patients with a history of alcohol or drug abuse in the last year
* Patients with a history of ischemic heart disease, peripheral artery disease, and/or cerebral vascular disease (including patients who have recently undergone coronary revascularization or angioplasty)
* Patients with a history of seizures, epileptic status and/or grand mal seizures
* History of chronic liver failure Child-Pugh A, B, and/or C
* History of acute renal failure (glomerular filtration rate <30 ml/min/1.72 m2)
* Patient with a history of chronic pain associated with fibromyalgia, Paget's disease or bone pain induced by metastatic cancer
* Low back pain due to a history of major trauma in the past 12 months (e.g., vertebral fracture, post-traumatic spondylolisthesis) or due to a visceral disorder (e.g., dysmenorrhea, history of endometriosis).
* Patients with symptoms suggestive of COVID-19 infection (fever, cough, dyspnea) and/or contact in the last 14 days with a suspected or positive patient for COVID-19

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients reporting pain improvement (reduction in pain intensity with a VAS ≤20 mm) at 1, 3, 5, and 7 days of follow-up, according to their baseline measurement in each treatment group | 7 dyas
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. At the end of the clinical trial the change porcentage will be measured and compared between treatment groups.
  The patient will visit the clinic at days 0,3 and 7. The researcher will call the patient for follow up at days 1 and 5.
Number of participants with treatment-related adverse events through the patient's diary record. | 7 dyas
  To describe the frequency, intensity and causality of the adverse events presented during the clinical trial by treatment group. The adverse events will be registered by the patient in the diary record. Each adverse event will be followed up at the discretion of the researcher.

SECONDARY OUTCOMES:
Analyze the average change in pain intensity according to VAS score at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. At the end of the clinical trial the change porcentage will be measured and compared between treatment groups.
  The patient will visit the clinic at days 0,3 and 7. The researcher will call the patient for follow up at days 1 and 5.
Analyze the percentage change in pain intensity based on VAS score at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  % change= ((Final Measurement-Initial Measurement)/(Initial Measurement))*100
Comparison of the proportion of subjects with pain improvement (reduction in pain intensity) through VAS, ≥ 30% at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. The proportion of patiens with an improvement of pain >30% will be reported and compared between treatment groups at days 1,3,5 and 7.
Comparison of the proportion of subjects with pain improvement (reduction in pain intensity) through VAS, ≥ 50% at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. The proportion of patiens with an improvement of pain >30% will be reported and compared between treatment groups at days 1,3,5 and 7.
Assess and compare the degree of physical disability due to acute low back pain, measured through the Oswestry disability questionnaire at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  The Oswestry questionnaire has been designed to give us information as to how the back pain has affected the ability to manage everyday life of patients, it classifies QOL as: no disability, mild disability, moderate disability, severe disability and completely disabled. The disability degree would be compared.
Assess and compare the degree of disability to perform daily activities due to low back pain, reported through Roland-Morris questionnaire at 1, 3, 5, and 7 days in each treatment group and in comparison with the baseline measurement. | 7 days
  The Roland-Morris questionnaire has been designed to assess the activities of daily living functional mobility pain. A maximum score of 24 indicates the greatest degree of disability from pain. The disability degree will be compared.
Assess changes in the score on the "Douleur Neuropathique-4 items" scale (DN-4) at days 3 and 7 in each treatment group and in comparison with the baseline measurement. | 7 days
  The DN4 is a clinician-administered, neuropathic pain diagnostic questionnaire, consisting of ten items grouped in four sections. The first seven items are related to the quality of pain (burning, painful cold, electric shocks) and its association to abnormal sensations (tingling, pins and needles, numbness, itching). The other three items are related to neurological examination in the painful area (touch hypoesthesia, pinprick hypoesthesia, tactile allodynia).
Report the number of patients who present therapeutic failure during the study among the treatment groups | 7 days
  Therapeutic failure will be defined by the principal researcher previous medical consult, the following criteria must be present:
  - When there is a decrease <10 mm or increase in VAS values compared to baseline and a ≥ 80% adherence to treatment

OTHER OUTCOMES:
To report the percentage of therapeutic adherence at day 7 of the intervention in each treatment group. | 7 days
  Therapeutic adherence will be defined by the principal researcher. Adherence to treatment will be defined as a consumption ≥ 80% of the doses that the patient should have ingested at the time of the corresponding evaluation.
Report the number of patients who require the use of rescue medication during the clinical trial in each treatment group | 7 days
  The rescue medication will be tramadol 50 mg:
  - The patient that considers the need for rescue medication must call the doctor, who will be in charge of applying the VAS scale by telephone. If the doctor considers it necessary, the taking of the rescue medication will be indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Choza-Romero, MD, Principal Investigator — Centro de Atención e Investigación Clínica S.C.; Adelfia Urenda-Quezada, MD, Principal Investigator — Servicios Avanzados de Investigación Médica Mediadvance S.C.; Isabel E Rucker Joerg, MD, Principal Investigator — Clinical Research Institute S.C.; Jesus H Mendoza-Ramírez, MD, Principal Investigator — Unidad Clínica de Bioequivalencia, S. de R.L. de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martina SD, Vesta KS, Ripley TL. Etoricoxib: a highly selective COX-2 inhibitor. Ann Pharmacother. 2005 May;39(5):854-62. doi: 10.1345/aph.1E543. Epub 2005 Apr 12. PMID 15827069
- [Background] Takemoto JK, Reynolds JK, Remsberg CM, Vega-Villa KR, Davies NM. Clinical pharmacokinetic and pharmacodynamic profile of etoricoxib. Clin Pharmacokinet. 2008;47(11):703-20. doi: 10.2165/00003088-200847110-00002. PMID 18840026
- [Background] Chiu CK, Low TH, Tey YS, Singh VA, Shong HK. The efficacy and safety of intramuscular injections of methylcobalamin in patients with chronic nonspecific low back pain: a randomised controlled trial. Singapore Med J. 2011 Dec;52(12):868-73. PMID 22159928
- [Background] Pallay RM, Seger W, Adler JL, Ettlinger RE, Quaidoo EA, Lipetz R, O'Brien K, Mucciola L, Skalky CS, Petruschke RA, Bohidar NR, Geba GP. Etoricoxib reduced pain and disability and improved quality of life in patients with chronic low back pain: a 3 month, randomized, controlled trial. Scand J Rheumatol. 2004;33(4):257-66. doi: 10.1080/03009740410005728. PMID 15370723
- [Background] Letizia Mauro G, Lauricella L, Vecchio M, Tomasello S, Scaturro D. Efficacy and tolerability of a fixed dose combination of cortex phospholipid liposomes and cyanocobalamin for intramuscular use in peripheral neuropathies. Minerva Med. 2019 Oct;110(5):455-463. doi: 10.23736/S0026-4806.19.06068-3. PMID 31368292
- [Background] Zhang YF, Ning G. Mecobalamin. Expert Opin Investig Drugs. 2008 Jun;17(6):953-64. doi: 10.1517/13543784.17.6.953. PMID 18491996
- [Background] Peracchi M, Bamonti Catena F, Pomati M, De Franceschi M, Scalabrino G. Human cobalamin deficiency: alterations in serum tumour necrosis factor-alpha and epidermal growth factor. Eur J Haematol. 2001 Aug;67(2):123-7. doi: 10.1034/j.1600-0609.2001.t01-1-00507.x. PMID 11722601
- [Background] Mauro GL, Martorana U, Cataldo P, Brancato G, Letizia G. Vitamin B12 in low back pain: a randomised, double-blind, placebo-controlled study. Eur Rev Med Pharmacol Sci. 2000 May-Jun;4(3):53-8. PMID 11558625
- [Background] Calderon-Ospina CA, Nava-Mesa MO, Arbelaez Ariza CE. Effect of Combined Diclofenac and B Vitamins (Thiamine, Pyridoxine, and Cyanocobalamin) for Low Back Pain Management: Systematic Review and Meta-analysis. Pain Med. 2020 Apr 1;21(4):766-781. doi: 10.1093/pm/pnz216. PMID 31529101
- [Background] Bacchi S, Palumbo P, Sponta A, Coppolino MF. Clinical pharmacology of non-steroidal anti-inflammatory drugs: a review. Antiinflamm Antiallergy Agents Med Chem. 2012;11(1):52-64. doi: 10.2174/187152312803476255. PMID 22934743
- [Background] Antoniou K, Malamas M, Drosos AA. Clinical pharmacology of celecoxib, a COX-2 selective inhibitor. Expert Opin Pharmacother. 2007 Aug;8(11):1719-32. doi: 10.1517/14656566.8.11.1719. PMID 17685888
- [Background] Smeets R, Koke A, Lin CW, Ferreira M, Demoulin C. Measures of function in low back pain/disorders: Low Back Pain Rating Scale (LBPRS), Oswestry Disability Index (ODI), Progressive Isoinertial Lifting Evaluation (PILE), Quebec Back Pain Disability Scale (QBPDS), and Roland-Morris Disability Questionnaire (RDQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S158-73. doi: 10.1002/acr.20542. No abstract available. PMID 22588742
- [Background] Shukla AK, Jhaj R, Misra S, Ahmed SN, Nanda M, Chaudhary D. Agreement between WHO-UMC causality scale and the Naranjo algorithm for causality assessment of adverse drug reactions. J Family Med Prim Care. 2021 Sep;10(9):3303-3308. doi: 10.4103/jfmpc.jfmpc_831_21. Epub 2021 Sep 30. PMID 34760748
- [Background] Mibielli MA, Geller M, Cohen JC, Goldberg SG, Cohen MT, Nunes CP, Oliveira LB, da Fonseca AS. Diclofenac plus B vitamins versus diclofenac monotherapy in lumbago: the DOLOR study. Curr Med Res Opin. 2009 Nov;25(11):2589-99. doi: 10.3111/13696990903246911. PMID 19731994